CLINICAL TRIAL: NCT05377047
Title: Treatment of Oligometastatic Breast Cancer - a Randomised Phase 3 Trial Comparing Stereotactic Ablative Radiotherapy and Systemic Treatment With Systemic Treatment Alone as 1st Line Treatment
Brief Title: Stereotactic Ablative Radiotherapy for OligoMetastatic Breast Cancer
Acronym: TAORMINA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Sahlgrenska University Hospital (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Region Örebro County (Other); Skane University Hospital (Other); Uppsala University Hospital (Other); Karolinska University Hospital (Other); University Hospital, Umeå (Other); Sundsvall Hospital (Other); Karlstad Central Hospital (Other); Gävle Hospital (Other); Centrallasarettet Västerås (Other); Oslo University Hospital (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); University of Stavanger (Other); University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SABO 21-01
Record Dates: First submitted 2022-04-11; First posted 2022-05-17 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer Stage IV; Oligometastatic Disease
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomisation 2:1 (systemic treatment + SABR vs systemic treatment)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental SABR arm (Experimental): Standard first line systemic therapy + SABR.
  Interventions: Radiation: SABR
- Control systemic therapy arm (No Intervention): Standard first line systemic therapy.

INTERVENTIONS:
Radiation: SABR — Stereotactic Ablative Radiotherapy is delivered to all metastatic lesions.
  Arms: Experimental SABR arm

SUMMARY:
TAORMINA is an international, multicentre, randomised phase 3 trial for patients with oligometastatic breast cancer (OMBC) that will be allocated to combined stereotactic ablative radiotherapy (SABR) + systemic therapy (investigational arm) versus systemic therapy alone (control arm) as 1st line therapy.

DETAILED DESCRIPTION:
TAORMINA is an international, multicentre, randomised phase 3 trial for patients with oligometastatic breast cancer (OMBC) that will be allocated to combined stereotactic ablative radiotherapy (SABR) + systemic therapy (investigational arm) versus systemic therapy alone (control arm) as 1st line therapy.

Patients with 1-5 metastases in 1-2 organs (confirmed by PET-CT) with any breast cancer subtype can be enrolled. All metastases must be available for SABR.

The primary aim is to investigate if the addition of SABR to the oligometastatic sites in addition to the standard first-line treatment can improve progression-free survival (PFS).

Secondary aims are to compare overall survival (OS), response rate and time to development of new lesions, acute and late toxicity. quality of life, time to start of chemotherapy (luminal patients).

Exploratory analyses:

Circulating tumour DNA as an early sign of disease progression. Immun panel for determination of the effect of SABR on patients´ immune response.

To investigate the survival for each BC subtype (Luminal, HER2+ and TNBC). To investigate survival in patients with de novo OMBC and recurrent OMBC respectively.

Stratifications are based on subtype (luminal, HER2-positive vs TNBC) and type of OMBC (de novo vs. recurrent) without formal sample size calculation for the stratification factor (exploratory analysis).

Patients with de novo metastatic OMBC that is planned for neoadjuvant treatment are recommended to complete treatment followed by standard surgery and radiotherapy or SABR towards the primary tumour lesion(s).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytological confirmed recurrent OMBC.
2. Age ≥18 years old.
3. OMBC defined as 1-5 metastases in a maximum of two organs confirmed by PET-CT.
4. Patients already on 1st line systemic treatment can be enrolled if repeated tumour evaluations show stable disease.
5. Patients with de novo stage IV OMBC must have a controlled primary tumour regardless of primary surgery or primary systemic treatment.
6. Patients with local recurrence and OMBC must have a controlled local recurrence.
7. ECOG/WHO 0-2.
8. Life expectancy > 6 months.
9. Known ER, PgR and HER2 status of either primary tumour or metastasis (preferred).
10. If measurable lesions, each ≤ 5 cm.
11. Symptomatic bone metastases are allowed if ablative therapy can be delivered (femoral metastasis not allowed).
12. Adequate organ function for the planned treatment according to local guide-lines.
13. For patients with liver metastasis:

    * No cirrhosis or hepatitis
    * Hepatic function:

      * Total bilirubin level < 3.0 x institutional ULN
      * ALT, AST, GGT, and alkaline phosphatase levels < 3.0 x institutional ULN
      * Albumin > 2.5 mg/dL
    * Metastasis not adjutant to stomach or small bowel.
14. For patients with abdominal metastases: adequate renal function with a calculated creatinine clearance of > 60mL/min.
15. Toxicities from previous adjuvant therapies (excluding alopecia) must have recovered to grade 1 (defined by CTCAE 5.0). Stable grade 2 peripheral neuropathy are considered individually by the investigator.
16. Negative pregnancy test within 14 days prior to start of treatment*.
17. If childbearing potential, willing to use an effective form of contraception*.
18. No other malignancy during the last 5 years except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix.
19. Signed informed consent and willingness to follow the trial procedures.

Exclusion Criteria:

1. > 1 line of systemic treatment for OMBC due to previous progressing disease (previous treatment of isolated local recurrences with a 2nd adjuvant treatment not included).
2. Oligometastases in brain.
3. Malignant pleural effusion or ascites.
4. Metastasis growth that involves > 3 vertebra and adjacent spinal cord, spine instability or neurological deficit resulting from compression, 25% spinal canal compromise or progressive neurological deficit.
5. Unable to undergo imaging by either CT scan or MRI.
6. Evidence of any other medical conditions (such as psychiatric illness, infectious diseases, neurological conditions, physical examination or laboratory findings) that may interfere with the planned treatment or affect patient compliance.
7. Pregnancy or breast-feeding.
8. Concurrent malignancy requiring therapy (excluding non-invasive carcinoma or carcinoma in situ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 years after the last patient inclusion
  Time from the date of randomisation to the date of disease-progression at any site or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years after the last patient inclusion
  Time from the date of randomisation to the date of death from any cause.
Local Control Rate (LCR) | 3 years after the last patient inclusion
  Time from the date of randomisation to the date of progress in previously treated metastases
Safety analysis - acute toxicity | From the first dose of SABR to 3 months after the last dose of SABR
  Reported according to CTCAE v.5.0
Safety analysis - late toxicity | From the first dose of SABR to 3 years after the last dose of SABR
  Reported according to CTCAE v.5.0
Health-related quality of life Cancer-30 | At base-line and after 3, 6, 9, 12, 18, 24 and 36 months after registration.
  European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaires Cancer-30 (EORTC-QLQ C30)
Health-related quality of life Breast-23 | At base-line and after 3, 6, 9, 12, 18, 24 and 36 months after registration.
  European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire Breast-23 (EORTC-QLQ B23)

CONTACTS AND LOCATIONS:
Overall Officials: Barbro K Linderholm, MD, PhD, Principal Investigator — Sahlgrenska University Hospital, Gothenburg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Milano MT, Zhang H, Metcalfe SK, Muhs AG, Okunieff P. Oligometastatic breast cancer treated with curative-intent stereotactic body radiation therapy. Breast Cancer Res Treat. 2009 Jun;115(3):601-8. doi: 10.1007/s10549-008-0157-4. Epub 2008 Aug 22. PMID 18719992
- [Result] Milano MT, Katz AW, Zhang H, Okunieff P. Oligometastases treated with stereotactic body radiotherapy: long-term follow-up of prospective study. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):878-86. doi: 10.1016/j.ijrobp.2011.08.036. Epub 2011 Dec 13. PMID 22172903
- [Result] Scorsetti M, Franceschini D, De Rose F, Comito T, Villa E, Iftode C, Navarria P, D'Agostino GR, Masci G, Torrisi R, Testori A, Tinterri C, Santoro A. Stereotactic body radiation therapy: A promising chance for oligometastatic breast cancer. Breast. 2016 Apr;26:11-7. doi: 10.1016/j.breast.2015.12.002. Epub 2016 Jan 3. PMID 27017237
- [Result] Milano MT, Katz AW, Zhang H, Huggins CF, Aujla KS, Okunieff P. Oligometastatic breast cancer treated with hypofractionated stereotactic radiotherapy: Some patients survive longer than a decade. Radiother Oncol. 2019 Feb;131:45-51. doi: 10.1016/j.radonc.2018.11.022. Epub 2018 Dec 28. PMID 30773186
- [Result] Trovo M, Furlan C, Polesel J, Fiorica F, Arcangeli S, Giaj-Levra N, Alongi F, Del Conte A, Militello L, Muraro E, Martorelli D, Spazzapan S, Berretta M. Radical radiation therapy for oligometastatic breast cancer: Results of a prospective phase II trial. Radiother Oncol. 2018 Jan;126(1):177-180. doi: 10.1016/j.radonc.2017.08.032. Epub 2017 Sep 21. PMID 28943046
- [Result] David S, Tan J, Savas P, Bressel M, Kelly D, Foroudi F, Loi S, Siva S. Stereotactic ablative body radiotherapy (SABR) for bone only oligometastatic breast cancer: A prospective clinical trial. Breast. 2020 Feb;49:55-62. doi: 10.1016/j.breast.2019.10.016. Epub 2019 Nov 6. PMID 31734589
- [Result] Li MP, Kelly D, Tan J, Siva S, Kron T, David S. Single-fraction stereotactic ablative body radiotherapy for sternal metastases in oligometastatic breast cancer: Technique and single institution experience. J Med Imaging Radiat Oncol. 2020 Aug;64(4):580-585. doi: 10.1111/1754-9485.13075. Epub 2020 Jun 25. PMID 32588550
- [Result] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754